CLINICAL TRIAL: NCT00093132
Title: A Phase 1/2 Study With Satraplatin and Simultaneous Radiation in Locally Advanced Non-Small Cell Lung Cancer
Brief Title: Satraplatin for Locally Advanced Non-Small Cell Lung Cancer With Simultaneous Radiotherapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decided to discontinue study drug development.
Sponsor: Agennix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAT1-04-02
Record Dates: First submitted 2004-10-01; First posted 2004-10-04 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Carcinoma, Non-small Cell Lung; Lung Cancer
Keywords: Non-Small Cell Lung Cancer (stage II or III); NSCLC; Squamous Cell Lung Cancer; adenocarcinoma of the lung; adenosquamous cell lung cancer; bronchoalveolar cell lung cancer; carcinoma, non-small cell lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — satraplatin

ARMS (1):
- Satraplatin (Experimental): Satraplatin
  Interventions: Drug: Satraplatin

INTERVENTIONS:
Drug: Satraplatin — Satraplatin is a member of the platinum-based class of chemotherapy drugs. Platinum-based drugs have been clinically proven to be one of the most effective classes of anticancer therapies. Unlike the currently marketed platinum-based drugs, satraplatin can be given orally.

SUMMARY:
PURPOSE: This trial is designed to compare the combination of the investigational oral cytotoxic drug, satraplatin, and radiation therapy for patients with locally advanced Non-Small Cell Lung Cancer (NSCLC) with no prior chemotherapy or radiation therapy treatment. Please refer to the Eligibility Criteria below for key inclusion and exclusion criteria.

WHAT IS SATRAPLATIN: Satraplatin is an oral, investigational anticancer drug that is a member of the platinum-based class of chemotherapy drugs. Platinum-based drugs have been clinically proven to be one of the most effective classes of anticancer therapies. Unlike the currently marketed platinum-based drugs, satraplatin can be given orally.

RATIONALE: Intravenously administered platinum-based drugs are currently used in combination with radiation therapy in the treatment of patients with locally advanced NSCLC. The purpose of this Phase I trial is to determine a tolerable dose and schedule for the oral platinum drug (satraplatin) when given to NSCLC patients throughout the course of their radiotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or medically inoperable NSCLC (stage II or III)
* ECOG performance status score 0-2
* Adequate bone marrow, liver, and pulmonary functions
* Life expectancy > three months.

Exclusion Criteria:

* Prior malignancy
* Serious concurrent uncontrolled medical disorder.
* Uncontrolled or significant cardiovascular disease
* History of mastectomy
* Pregnant or breast-feeding patients are not eligible
* Prior radiotherapy to the primary tumor site or cytotoxic chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-08; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Determination of MTD and recommended dose for phase II trials | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Southwestern Medical Center, Dallas, Texas, United States